CLINICAL TRIAL: NCT06495099
Title: Effect of Core Stability Exercises and Russian Electrical Stimulation in Non-specific Low Back Pain (Randomized Control Trail)
Brief Title: Effect of Core Stability Exercises and Russian Electrical Stimulation in Non-specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: physio 224
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): The training group A will be treated by core stability exercises and Russian electrical stimulation
  Interventions: Other: Russian electrical stimulation
- group B (Active Comparator): The training group B will be treated by core stability exercises.
  Interventions: Other: Russian electrical stimulation

INTERVENTIONS:
Other: Russian electrical stimulation — Type of Medium frequency current with 2500 Hz frequency modulated at 50 Hz with 50% Duty cycle training protocol is (10 sec. on time - 50 sec. off time - 10 minutes total time)

SUMMARY:
Brief Summary: Low back pain (LBP) is an important public health problem due to the increasing world population and aging. In chronic LBP, exercise therapy is among the first-line treatments. Core stabilization exercises (CSE), one of the motor control exercises, focus on the activation and control of the deep spinal muscles. Recently, some studies have shown that Russian electrical stimulation alone or combined with exercise can provide contraction in deep stabilizer muscles and significantly reduce pain in patients with LBP

ELIGIBILITY:
Inclusion Criteria:

* The duration of the disease is more than 3 months with pain scores greater than four in the VAS disability score of 19% or greater as evident from the modified oswestry disability.

Exclusion Criteria:

* Neurological or musculoskeletal diseases that affect lumbar spine (e.g: lumbar spondylosis, spondylolisthesis, and lumbar disc injuries)
* women during pregnancy and lactation.
* History of lumbar spine surgery.
* Signs of lumbar radiculopathy or myelopathy.
* Signs of serious pathology (e.g., malignancy, inflammatory disorders, infection

Ages: 20 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Pain scoring | 6 weeks
  pain measured by VAS tool, 0 the least pain while 10 the highest one
Quality of life by using Oswestry Disability Index (OID) | 6 weeks
  questioner, Score from 0 to 19% indicate minimal disability- 20 to 39% represent moderate disability- 40 to 59% represent severe disability- 60 to 79% represent crippled disability- and scores from 80 to 100% represents patients that are confined to bed

SECONDARY OUTCOMES:
Muscle thickness assessment | 6 weeks
  Ultrasonography
Stability and mobility of spine | 6 weeks
  Spinal mouse assessment spinal vertebrate from 7th cervical vertebrae to 3rd sacral vertebrae

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No